CLINICAL TRIAL: NCT07130396
Title: A Single Arm Trial to Evaluate the Effect of PhytoMulti® Multivitamin and UltraFlora® Balance Probiotic on Bowel Symptoms in Individuals Using GLP-1 Receptor Agonists, Assessed by the IBS Symptom Severity Score (IBS-SSS)
Brief Title: Impact of Multivitamin (PhytoMulti®) and a Probiotic (UltraFlora® Balance Probiotic) on Gut Health of People Taking GLP-1 Medication
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Metagenics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: GLO-NAM-2025-02
Record Dates: First submitted 2025-08-12; First posted 2025-08-19 (Actual); Last update posted 2025-08-19 (Actual); Status verified 2025-08

CONDITIONS: GLP-1; Adults
MeSH Terms: interventions — Geritol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- PhytoMulti® Multivitamin and UltraFlora® Balance Probiotic arm (Active Comparator)
  Interventions: Dietary Supplement: Multivitamin and a Probiotic

INTERVENTIONS:
Dietary Supplement: Multivitamin and a Probiotic — The duration of trial intervention and participation for an individual participant is approximately 3 months (12 weeks). Screening, during which eligibility to participate in the trial is assessed, occurs at baseline. A fixed, orally administered, dose of the study products (PhytoMulti® Multivitamin, 2 tablets/day and UltraFlora® Balance Probiotic, 1 capsule/day) are taken daily with breakfast

SUMMARY:
This is a single-arm, open-label clinical trial involving 100 participants who will undergo a total participation period of 12 weeks.

DETAILED DESCRIPTION:
The trial begins with a screening to assess eligibility, followed by a 12-week treatment phase during which participants will receive a fixed-dose oral supplementation regimen. During this treatment period, participants will take PhytoMulti® Multivitamin at a fixed dose of 2 tablets per day and UltraFlora® Balance Probiotic at a fixed dose of 1 capsule per day, both administered orally once daily with food. During the 12-week treatment period, participants will be asked to complete questions at fixed timepoints.

ELIGIBILITY:
Inclusion Criteria:

1. Providing written informed consent
2. Males and females of at least 18 years old
3. Minimum 4 weeks on GLP-1 (f.e Ozempic®, Wegovy®, Mounjaro®, etc.) and maximum 1 year on GLP-1
4. Body Mass Index (BMI) ≥ 25 AND ≤ 30
5. Being willing to maintain stable dietary habits and physical activity levels throughout the trial period
6. Being willing not to introduce any other food supplements during the trial period (supplements used in the two weeks prior to enrolling in the trial and used consistently throughout are acceptable, except for probiotics).

Exclusion Criteria:

1. Having had any type of bariatric surgery, or planned bariatric surgery during the period of trial participation.
2. Suffering from a severe chronic disease (e.g., cancer, HIV, hepatic or renal impairment, diabetes type I), inflammatory bowel disease (IBD), Coeliac Disease, and/or being immunocompromised.
3. Suffering from any uncontrolled endocrine disorder
4. Having used any antibiotic treatment in the 2 months prior to enrollment.
5. Having a known allergy to the ingredients in the study product.
6. Being pregnant or lactating (breastfeeding) or trying to become pregnant.
7. Participating in another clinical trial.
8. Suffering from dementia or inability to take the trial treatment in an appropriate way.
9. Taking PhytoMulti® Multivitamin and/or UltraFlora® Probiotic or any similar product from competitors prior to trial participation

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2025-11-01 (Estimated); Primary Completion 2026-03-31 (Estimated); Study Completion 2026-04-30 (Estimated)

PRIMARY OUTCOMES:
IBS- SSS | From enrollment to the end of treatment at 12 weeks (90 days)
  To assess impact of PhytoMulti® multivitamin and UltraFlora® Balance Probiotic on abdominal symptoms using the IBS severity scoring system (IBS-SSS)

CONTACTS AND LOCATIONS:
Overall Officials: Mieke Van Den Driessche, PhD, Study Director — Metagenics, Inc.; Irfan Qureshi, MD, Principal Investigator — Metagenics, Inc.

IPD SHARING:
Plan to Share IPD: No